CLINICAL TRIAL: NCT06540274
Title: Outcomes and Complications of Surgery for Degenerative Lumbar Spine Diseases in Elderly Patients Above 65 Years.
Brief Title: Outcomes of Surgery for Degenerative Lumbar Spine Diseases
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohammed Zaki Morsi, Director, Assiut University
Other Study IDs: Lumbar spine surgery in elders
Record Dates: First submitted 2024-06-10; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Degenerative Lumbar Spine Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: lumbar surgery — Discectomy, lumbar fusion or laminectomy

SUMMARY:
The purpose of this study is to determine the effectiveness of surgery on the elderly patients with DSD.

DETAILED DESCRIPTION:
This study based on observation and follow up of elderly patients underwent for surgery for degenrtative lumbar spine diseases and the effectiveness of the surgery on the quality of their life.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders with age above 65 years with Low Back Pain and disability.
* Pt with clinical diagnosis of degenerative lumbar spine disease.
* Pt with MRI showing Degenerative lumbar spine disease need surgical intervention.

Exclusion Criteria:

* Patients having malignancy, vertebral fractures, trauma, inflammatory illnesses, and infection.
* Patients with degenerative conditions in the cervical and /or thoracic spine.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: The study on the elderly patients of both genders with degenerative lumbar spine diseases.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale (VAS). | baseline
  Subjective measurement for back and leg pain.The highest degree which consider worse is 8-10 and the degree which consider better is 0-3

SECONDARY OUTCOMES:
Oswestry Disability Index. | baseline
  To measure satisfaction of the patient and the functional disability. The score 0-20 consider better and the score 40-100 consider worse

CONTACTS AND LOCATIONS:
Locations (1):
- Mahmoud, Asyut, Egypt